CLINICAL TRIAL: NCT02287740
Title: Comparative Effectiveness and Cost-effectiveness of a Fall Prevention Intervention: Tai Ji Quan: Moving for Better Balance
Brief Title: Prevention of Falls Among Older Adults in Community Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AG045094-01A1 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-11-11 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Fall
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tai Ji Quan: Moving for Better Balance (Experimental): This protocol involves training 2 times a week for 6 months.
  Interventions: Behavioral: Tai Ji Quan: Moving for Better Balance
- Multimodal Exercise (Active Comparator): This protocol involves training 2 times a week for 6 months.
  Interventions: Behavioral: Multimodal Exercise
- Stretching (Sham Comparator): This protocol involves participation of 2 times a week for 6 months.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Tai Ji Quan: Moving for Better Balance — The protocol involves a core 8-form routine training with built-in variations and a subroutine of integrated therapeutic movements.
  Arms: Tai Ji Quan: Moving for Better Balance
Behavioral: Multimodal Exercise — The protocol involves a multi-modality program that involves aerobic, strength, balance, and flexibility exercises.
  Arms: Multimodal Exercise
Behavioral: Stretching — The protocol represents a minimum standard of practice for exercises for older adults with activities consisting primarily of seated exercises accompanied by breathing, stretching, and relaxation.
  Arms: Stretching

SUMMARY:
Objective: To conduct a comparative efficacy and cost-effectiveness study of an evidence-based fall prevention program-Tai Ji Quan: Moving for Better Balance (TJQMBB).

DETAILED DESCRIPTION:
To determine the effectiveness and cost-effectiveness of the two evidence-based exercise programs (Multimodal Exercise,TJQMBB) relative to stretching, a proxy for a minimum practice standard, in reducing falls among older adults at risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* aged 70 years or older living independently in the community
* at least one fall in the preceding 12 months and a referral from a healthcare provider indicating the participant is at risk of falls due to gait/balance impairment or medication use or impaired mobility as evidenced by Timed Up and Go result of >13.5 seconds
* no participation in daily and/or structured vigorous physical activity or walking for exercise that lasted 15 minutes or longer at a time or muscle-strengthening activities on 2 or more days a week in the previous 3 months
* walking independently, with or without the use of an assistive device,
* no severe cognitive impairment (Mini-Mental State Examination score ≥20)
* able to exercise safely as determined by their healthcare provider,
* a willingness to be randomly assigned to an intervention condition and complete the 6-month intervention and 6 month follow-up.

Exclusion Criteria:

* any medical or physical conditions deemed unacceptable by their physician or healthcare provider,
* planned to leave the study area within the next 12 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 670 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the number of falls | Baseline, 6 Months
  Using a daily diary "fall calendar," falls reported by participants across the 24-week surveillance period will be collected, starting from the date of first intervention class and continuing until participants withdrew, had died or were lost to follow-up.

SECONDARY OUTCOMES:
Functional Reach | Baseline, 6 Months
  assessing the maximal distance (in inch) participants one can reach forward, beyond arm's length, while maintaining a fixed based of support in the standing position. Differences between baseline and 6 months scores will be calculated to assess change.
Instrumented Timed Up and Go | Baseline, 6 Months
  assessing the time to complete a series of functional tasks (sit-to-stand, 180 degree turn, turn-to-sit.) while walking through a 7-meter walkway (7 meters towards a line, turn, and 7 meters towards the chair). The measure is assessed in second. Differences between baseline and 6 months scores will be calculated to assess change.
Physical Performance | Baseline, 6 Months
  The physical performance measure consists of 4-meter walk at usual pace, a timed repeated chair stand, and 3 increasingly difficult standing balance tests. Each measure is assigned a categorical score ranging from 0 (inability to complete the test) to 4 (best performance). A summary score ranging from 0 (worst performance) to 12 (best performances) will be calculated by summing the 3 components scores.
Cognitive function | Baseline, 6 Months
  Montreal Cognitive Assessment (in points). Differences between baseline and 6 months scores will be calculated to assess change.
Cost per fall prevented | Baseline, 6 Months
  determined by calculating total intervention cost estimates divided by number of falls observed during the 6 month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhong Li, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Li F, Harmer P, Eckstrom E, Fitzgerald K, Chou LS, Liu Y. Effectiveness of Tai Ji Quan vs Multimodal and Stretching Exercise Interventions for Reducing Injurious Falls in Older Adults at High Risk of Falling: Follow-up Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2019 Feb 1;2(2):e188280. doi: 10.1001/jamanetworkopen.2018.8280. PMID 30768195
- [Derived] Li F, Harmer P, Eckstrom E, Fitzgerald K, Akers L, Chou LS, Pidgeon D, Voit J, Winters-Stone K. Cost-Effectiveness of a Therapeutic Tai Ji Quan Fall Prevention Intervention for Older Adults at High Risk of Falling. J Gerontol A Biol Sci Med Sci. 2019 Aug 16;74(9):1504-1510. doi: 10.1093/gerona/glz008. PMID 30629121
- [Derived] Li F, Harmer P, Fitzgerald K, Eckstrom E, Akers L, Chou LS, Pidgeon D, Voit J, Winters-Stone K. Effectiveness of a Therapeutic Tai Ji Quan Intervention vs a Multimodal Exercise Intervention to Prevent Falls Among Older Adults at High Risk of Falling: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1301-1310. doi: 10.1001/jamainternmed.2018.3915. PMID 30208396